CLINICAL TRIAL: NCT06236360
Title: The Effect of Individualized Nutritive Intervention Based on the Mediterranean Diet on the Changes in the Gut Microbiome, Quality of Life, and Radiological and Biochemical Response to Immunotherapy in Metastatic Melanoma Patients
Brief Title: Metastatic Melanoma Patients on Immunotherapy With Nutritive Intervention Based on Mediterranean Diet
Acronym: MINI-MD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Rijeka (Other)
Responsible Party: Principal Investigator, Marin Golčić, Deputy lead investigator, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 8.1-23/262-6
Record Dates: First submitted 2023-12-21; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Melanoma Stage Iv; Metastatic Melanoma
Keywords: melanoma; immunotherapy; metastasis; mediterranean diet
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators/care providers will be masked, while investigators performing nutritional interventions will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet intervention (Experimental): The intervention study will involve scheduled communications (via phone, video call, and/or email) with a trained nutritionist based on protocol-determined parameters and recommendations, organized weekly in the first month, every other week in the second month, and once a month in the third month. Each patient will receive general guidance and information about the MD. Additionally, a personalized nutritional plan based on the MD will be prepared for each patient, considering their initial dietary habits, preferences, food accessibility, and financial constraints. Throughout the 12-week period, patients will be motivated to adhere to the prescribed dietary regimen.
  Interventions: Behavioral: Mediterranean Diet Intervention
- Continuing with previous diet (No Intervention): The control group will continue with their usual/current diet, with the exception of supplementation of those in whom low serum vitamin D level (in accordance with current medical recommendations)

INTERVENTIONS:
Behavioral: Mediterranean Diet Intervention — The primary goal is to evaluate whether tele-intervention can elevate the level of flavonoids, anthocyanins, proteins, omega-3 fatty acids, short fatty acids, fruits and vegetables, and fibers (all previously associated with a better response to immunotherapy) and limit foods with added sugars.
  Arms: Mediterranean diet intervention

SUMMARY:
This research will study the effect of Mediterranean diet intervention in patients undergoing immunotherapy treatment for metastatic melanoma and its relationship with gut microbiome and quality of life. One group of patients will continue with their regular diet, while the other will receive dietary tele-intervention with trained nutritionist during the 12-week period. Gut microbiome, quality of life questionnaires, blood parameters and radiological examination will be evaluated before and 12-weeks after the start of the intervention.

DETAILED DESCRIPTION:
Metastatic melanoma is a malignant tumor of melanocyte origin that has spread to other organs. The basis of treatment is systemic therapy, most commonly anti-programmed death-1 (PD-1) and anti- cytotoxic T-lymphocyte-associated protein 4 (CTLA- 4) immunotherapy, although for some patients, thyrosine kinase inhibition is also a treatment option. Survival of metastatic melanoma patients has been significantly extended over the last decade, and the use of immunotherapy has led to a median overall survival of 72 months and a response rate of up to 60%. However, not all cancer patients respond equally to immunotherapy, and the variation in response may be attributed to the individual's microbiome, which is heavily influenced by dietary habits. Over 2/3 of patients will progress during the 6.5 years of follow-up and currently there is a limited number prognostic and predictive parameters to assess the response to immunotherapy. However, understanding and manipulating the microbiome through dietary interventions offers a potential avenue for enhancing immunotherapy outcomes in cancer patients and, consequently, may serve as a complementary therapeutic strategy. Due to previous data, as well as investigators' previous publication on the importance of gut microbiome as a co-denominator for immunotherapy response, and aiming towards constructing a protocol on dietary intervention for enhancing immunotherapy response in metastatic melanoma patients, the investigators evaluated a systematic search for the data showing association with an improved immunotherapy response.

A diet with moderately elevated sodium use (2.3-4 g daily), diet rich in fiber (20-25 g daily), fruits and vegetables (≥5 servings daily), vitamin D, 23 omega-3 fatty acids and whole grains (≥3 servings daily) has been associated with a more diverse and beneficial microbiome, which in turn promotes the production of short-chain fatty acids (SCFA). All the listed foods belong to the Mediterranean diet (MD), which is based on fresh fruits and vegetables, legumes, olive oil, and unrefined fiber. MD also includes a lower intake of meat, eggs, processed foods, sugars, and saturated fatty acids, which may all lead to a less diverse and potentially less favorable microbiome and health outcomes. Various clinical studies already demonstrated the beneficial effect of MD in non-oncology patients. As for oncology patients, the benefit of the MD in reducing the incidence of cancer has been known for many years, especially for breast cancer patients. Furthermore, a published cohort study with 52 patients receiving immune checkpoint blockade (ICB) treatment for various solid tumors revealed that higher fecal SCFA concentrations were associated with longer progression-free survival. Another cohort study comprising patients with advanced melanoma in the UK and the Netherlands, demonstrated that a stronger adherence to the MD principles was linked to a higher likelihood of responding positively to ICB treatment. However, there is a scarcity of randomized trials evaluating the effect of the nutritional intervention based on the MD in cancer patients undergoing treatment. As far as the investigators are aware, there are no current clinical trials applying a nutritional intervention based on the MD in patients with metastatic melanoma; however, there is an ongoing randomized DIET study - NCT04645680 (with expected ending in 2024), aiming to evaluate effectiveness of fiber-enriched diet within the melanoma setting. The potential effect of the MD based nutritional intervention could result in a greater benefit compared to trials focusing only on one nutrient. Considering the issues learned from COVID-19 pandemic, the main goal of the trial is to determine the effectiveness and applicability of a remote personalized nutritional intervention based on the MD to increase the intake of micronutrients (flavones, anthocyanins, omega-3 fatty acids, vitamin D and fiber) previously associated with a positive response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* pathophysiologically confirmed cutaneous melanoma stage IV or inoperable stage IIIC,
* radiologically measurable disease on computerized tomography (CT) or positron emission tomography (PET)/CT,
* The multidisciplinary team recommended initiation of treatment with dual immunotherapy with anti-PD-1 + anti-CTLA4 immunotherapy
* written informed consent prior to participation
* willingness to monitor and adjust the dietary regimen if necessary
* Eastern Cooperative Oncology Group (ECOG) status 0-1.

Exclusion Criteria:

* lifetime history of psychiatric disorders
* active brain metastases
* active autoimmune disease
* systemic use of equal or more than 10 mg of prednisone or an appropriate corticosteroid equivalent during screening
* exposure to antibiotics and probiotics or other supplements that can affect the study outcome during screening within the last 3 weeks,
* uncontrolled diabetes
* history of clinically significant drug or alcohol abuse within the last 6 months
* specific dietary habits that are not inclined or able to change or the existence of food allergy or intolerance to certain food
* inability or refusal to participate in all research procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the level of ingested flavones | From enrollment to the end of treatment at 12 weeks
  To evaluate the effectiveness and applicability of a tele-individualized nutritional intervention based on the Mediterranean diet (INIMP) to increase the intake of micronutrients (flavones)
Change in the level of ingested anthocyanins | From enrollment to the end of treatment at 12 weeks
  To evaluate the effectiveness and applicability of a tele-individualized nutritional intervention based on the Mediterranean diet (INIMP) to increase the intake of micronutrients (anthocyanin)
Change in the level of ingested omega-3 fatty acids | From enrollment to the end of treatment at 12 weeks
  To evaluate the effectiveness and applicability of a tele-individualized nutritional intervention based on the Mediterranean diet (INIMP) to increase the intake of micronutrients (omega-3 fatty acids)
Change in the level of ingested vitamin D | From enrollment to the end of treatment at 12 weeks
  To evaluate the effectiveness and applicability of a tele-individualized nutritional intervention based on the Mediterranean diet (INIMP) to increase the intake of micronutrients (vitamin D)
Change in the level of ingested fibre | From enrollment to the end of treatment at 12 weeks
  To evaluate the effectiveness and applicability of a tele-individualized nutritional intervention based on the Mediterranean diet (INIMP) to increase the intake of micronutrients (fibre)

SECONDARY OUTCOMES:
A change in radiological response rate (PET/CT or CT) | From enrollment to the end of treatment at 12 weeks
  Assess the impact of INIMP on the radiological response rate (PET/CT or CT)
A change in gut microbiome strains associated with an improved response to immunotherapy | From enrollment to the end of treatment at 12 weeks
  Assess the impact of INIMP on changes in the microbiome
A change in the quality of life assessed by EORTC QLQ C15-PAL | From enrollment to the end of treatment at 12 weeks
  Assess the impact of INIMP on the quality of life measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 Palliative scores (EORTC QLQ-C15-PAL), which is a 'core questionnaire' for palliative care, measuring symptom burden and quality of life
A change of biochemical biomarkers of melanoma (S100 and LDH) | From enrollment to the end of treatment at 12 weeks
  Assess the impact of INIMP on biochemical biomarkers of melanoma (S100 and LDH)

OTHER OUTCOMES:
A change of concentration of microbiome associated with a good immune response | From enrollment to the end of treatment at 12 weeks
  evaluate the connection between changes in the intake of micronutrients and the microbiome
A correlation between microbiome associated with a good immune response and response | From enrollment to the end of treatment at 12 weeks
  To evaluate the association of the basic microbiome and the rate of biochemical and radiological response
A correlation between microbiome associated with a good immune response and less adverse effects | From enrollment to the end of treatment at 12 weeks
  To assess the association between the basic microbiome and the rate of immunotherapy side effects

CONTACTS AND LOCATIONS:
Overall Officials: Davorin Herceg, MD, PhD, Principal Investigator — CHC Zagreb
Locations (1):
- University Hospital Zagreb-Rebro, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data regarding the basic information and microbiome.
Supporting Information: Study Protocol, SAP
Time Frame: after 3 months from study termination up to 12 months later
Access Criteria: Following an official claim and review by a local Ethics Committee